CLINICAL TRIAL: NCT00232856
Title: A Multi-Center, Non-Randomised Study of the CYPHER™ Sirolimus-Eluting Stent in the Treatment of Patient With an in-Stent Restenotic Native Coronary Artery Lesion
Brief Title: A Study of the Cypher SES to Treat Restenotic Native Coronary Artery Lesions.
Acronym: TROPICAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Hans-Peter Stoll - Director Medical Affairs, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC01-06
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Cypher™ sirolimus-eluting stent
  Interventions: Device: drug-eluting stent

INTERVENTIONS:
Device: drug-eluting stent — PCI
  Other Names: Cypher™ sirolimus-eluting stent

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the Cypher™ sirolimus-eluting stent in reducing angiographic in-lesion late loss in patients with an in-stent restenotic native coronary artery lesion.

DETAILED DESCRIPTION:
This is a multicenter (11 sites), non-randomized study. Patients who meet the eligibility criteria will be treated with the Cypher™ sirolimus-eluting stent. All patients will have a repeat angiography at six months post-procedure and will be additionally followed clinically at 1, 6 and 9 months and up to 3 years. The results of this study will be compared with the outcome of the GAMMA I / II as the historical control.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has an in-stent restenosis of ≥ 60% and < 100% (by QCA online of the MLD compared to the distal reference diameter) in a native coronary artery.
2. The study target lesion can not be located in a vessel containing another lesion requiring treatment. Lesions located in other vessels may be treated with percutaneous revascularization at the time of the procedure, BUT they must be successfully treated prior to the treatment of the study target lesion.

Exclusion Criteria:

1. Unprotected left main coronary disease with ≥ 50% stenosis;
2. Patient previously treated with brachytherapy in any coronary vessel.
3. Target lesion involves bifurcation including a side branch >2.5mm in diameter.
4. The patient sustained a recent (<72 hours) myocardial infarction defined as a serum CK 2x the upper limit of normal and elevated MB or abnormal lab values.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2002-12; Primary Completion 2003-12 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
angiographic in-lesion late loss | 6 months post-procedure

SECONDARY OUTCOMES:
in-stent mean percent diameter stenosis (%DS) | 6-months post-procedure
i-stent late loss (LL) | 6 months post-procedure
in-lesion binary restenosis | 6-months post-procedure
Target Vessel Revascularization (TVR) | 9-months post-procedure
Target Vessel Failure (TVF) defined as any revascularization of the index vessel or myocardial infarction or death that cannot be clearly attributed to a vessel other than the index vessel | 9 months post-procedure
Composite of Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target lesion revascularization in-hospital | 1, 6, 9 months and, 2 and 3 years post-procedure
occurrence of bleeding | 1, 6, 9 months and, 2 and 3 years post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Franz-Josef Neumann, MD, Principal Investigator — Herz-zentrum Bad Krozingen; Walter Desmet, MD, Principal Investigator — K.U. Leuven
Locations (2):
- K.U. Leuven, Leuven, Belgium
- Herz-zentrum Bad Krozingen, Bad Krozingen, Germany